CLINICAL TRIAL: NCT01110759
Title: Retrospective Chart-review Study Involving Outpatients Who Underwent Hand Surgery With Local Anesthesia: Comparing Outcome With a Peripheral Nerve Block vs. Local Infiltration Alone
Brief Title: Medical Review: Hand Surgery After Local Block Versus Non-block
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ronald Wender, Chairman, Department of Anesthesiology, Cedars-Sinai Medical Center
Other Study IDs: Pro00019315
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: pain management; ambulatory surgery; opioid; local anesthesia; hand surgery; postoperative pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Agnosia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Under Local Infiltration
- Under Peripheral Nerve Block

SUMMARY:
In this study, the effects of local block vs non block will be assessed with respect to postoperative outcomes (such as pain score, and recovery profiles) in outpatients after hand surgery.

DETAILED DESCRIPTION:
Analyzing medical records and through a telephone questionnaire, in a retrospective and prospective review respectively.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Outpatients who underwent hand surgery under peripheral nerve block or local infiltration alone

Exclusion Criteria:

* Patients who do not meet inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients undergoing hand surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
postoperative pain | hours to months
  1. Severity of the pain experienced before patient left the surgery center and after patient arrived at home
  2. Pain medication (amounts of opioids and non opioids pills) required
  d)Time to suffer pain at the surgical site (hand) (days, weeks, or months)

SECONDARY OUTCOMES:
Nausea | days to weeks
  1. Severity of the nausea experienced by the patient.
  2. Medication required.
  3. Time to suffer nausea.
Vomiting | dias to weeks
  1. Severity
  2. Medication required
  3. Time to suffer vomiting

OTHER OUTCOMES:
Outcomes | days to weeks
  * Presence of any other problems: (e.g., headaches, dizziness, drowsiness, fatigue, constipation, difficulty voiding.)
  * Time taken to return to normal activities after surgery
  * Satisfaction with the pain management after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Wender, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States